CLINICAL TRIAL: NCT01085786
Title: Comparison of 14-day Sequential and Hybrid Therapies for H Pylori Infection
Brief Title: Sequential and Hybrid Therapies for H Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Baylor College of Medicine (Other); Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS97-CT6-08
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori infection
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 14-day sequential treatment (Active Comparator): One in which the first component consists of a proton pump inhibitor and amoxicillin given for 7 days followed by the PPI, clarithromycin and metronidazole for 7 days.
  Interventions: Drug: 14-day sequential treatment
- 14-day hybrid treatment (Experimental): esomeprazole 40 mg and amoxicillin 1 g twice daily for 7 days followed by esomeprazole 40 mg, amoxicillin 1 g, clarithromycin 500 mg and metronidazole 500 mg twice daily for 7 days
  Interventions: Drug: 14-day hybrid treatment

INTERVENTIONS:
Drug: 14-day sequential treatment — * 14-day sequential therapy arm: esomeprazole 40 mg and amoxicillin 1 g twice daily for 7 days followed by esomeprazole 40 mg, clarithromycin 500 mg and metronidazole 500 mg twice daily for 7 days
  * 14-day hybrid therapy arm: esomeprazole 40 mg and amoxicillin 1 g twice daily for 7 days followed by esomeprazole 40 mg, amoxicillin 1 g, clarithromycin 500 mg and metronidazole 500 mg twice daily for 7 days
  Other Names: Esomeprazole, amoxicillin, clarithromycin, metronidazole
  Arms: 14-day sequential treatment
Drug: 14-day hybrid treatment — esomeprazole 40 mg and amoxicillin 1 g twice daily for 7 days followed by esomeprazole 40 mg, amoxicillin 1 g, clarithromycin 500 mg and metronidazole 500 mg twice daily for 7 days
  Other Names: esomeprazole + amoxicillin, then quadruple therapy
  Arms: 14-day hybrid treatment

SUMMARY:
Primary: To evaluate efficacy of 14 day 2-phase sequential therapy given in two forms. One in which the first component consists of a proton pump inhibitor and amoxicillin given for 7 days followed by the PPI, clarithromycin and metronidazole for 7 days. The alternate will be similar with the exception that the amoxicillin will be continued throughout the 14 days. The secondary endpoint is to evaluate the effectiveness of therapy in relation to antibiotic resistance.

DETAILED DESCRIPTION:
The purpose of this study is to test whether the 14-day sequential therapy ( esomeprazole plus amoxicillin dual therapy for 7 days followed by triple therapy with esomeprazole, clarithromycin, and metronidazole for 7 days) or 14-day hybird therapy (esomeprazole plus amoxicillin dual therapy for 7 days followed by quadruple therapy with esomeprazole, amoxicillin, clarithromycin, and metronidazole for 7 days) can achieve an eradication rate equal to or more than 95%.

A total of 240 subjects will be asked to participate in this study.

H. pylori-infected patients are randomized to either a 14-day sequential therapy (esomeprazole 40 mg and amoxicillin 1 g twice daily for 7 days followed by esomeprazole 40 mg, clarithromycin 500 mg and metronidazole 500 mg twice daily for 7 days) or a hybrid therapy (esomeprazole 40 mg and amoxicillin 1 g twice daily for 7 days followed by esomeprazole 40 mg, amoxicillin 1 g, clarithromycin 500 mg and metronidazole 500 mg twice daily for 7 days).

Eradication efficacy is assessed by a follow-up endoscopy with rapid urease test and histological examination eight weeks after the end of anti-H. pylori therapy. The eradication rates of the two study groups will be compared.

A successful regimen is defined as a regimen achieving an eradication rate equal to or more than 95%.

ELIGIBILITY:
Inclusion Criteria:

* consecutive H. pylori-infected outpatients, at least 18 years of age, with endoscopically proven peptic ulcer diseases or gastritis

Exclusion Criteria:

* previous H. pylori-eradication therapy
* ingestion of antibiotics, bismuth, or PPIs within the prior 4 weeks
* patients with allergic history to the medications used
* patients with previous gastric surgery
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
* pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwok-Hung Lai, PhD, Study Chair — Kaohsiung Veterans General Hospital.; David Y Graham, MD, Study Director — Baylor College of Medicine; PING-I Hsu, MD, PhD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (2):
- Taiwan (2):
  - Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan
  - Kaohsiung Veterans General Hospital, Kaohsiung City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: Aug 2008 - May 2010
Pre-assignment Details: no significant events for the overall study
Period: Overall Study
Arm/Group | 14-day Sequential Treatment | 14-day Hybrid Treatment
Started | 123 | 117
Completed | 123 | 117
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 14-day Sequential Treatment | 14-day Hybrid Treatment | Total
Number analyzed (Participants) | 123 | 117 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 91 | 188
  >=65 years | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (11.8) | 54.3 (11.4) | 54.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 58 | 120
  Male | 61 | 59 | 120
Region of Enrollment [Number; unit: participants]
  Taiwan | 123 | 117 | 240

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Which H. Pylori Was Eradicated
Description: evaluate eradication outcome by endoscopy with urease test or urea breath test
Time Frame: Dec 2010
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | 14-day Sequential Treatment | 14-day Hybrid Treatment
Number analyzed (Participants) | 123 | 117
participants | 94 [90 to 98] | 99 [95 to 100]

2. Secondary Outcome: Adverse Events
Description: by standardized questionnaire
Time Frame: Dec 2010
Reporting Status: Not Posted
Measure: Number; unit: participants

3. Secondary Outcome: Compliance Rate
Description: Good compliance is defined as taking equal or more than 90% of eradication medicines
Time Frame: Dec 2010
Reporting Status: Not Posted
Measure: Number (95% Confidence Interval); unit: participant

ADVERSE EVENTS:
Time Frame: period of data collection: 12 months
Arm/Group | 14-day Sequential Treatment | 14-day Hybrid Treatment
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/117
Other Adverse Events (participants affected / at risk) | 26/123 | 17/117
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 14-day Sequential Treatment (N=123) | 14-day Hybrid Treatment (N=117)
Taste perversion (Gastrointestinal disorders) | 11 (11) | 8 (8)
nausea (Gastrointestinal disorders) | 13 (13) | 3 (3)
diarrhea (Gastrointestinal disorders) | 4 (4) | 8 (8)

LIMITATIONS AND CAVEATS:
The trial was performed in a single country.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes